CLINICAL TRIAL: NCT01380691
Title: A Study to Investigate the Pharmacodynamic and Pharmacokinetic Interaction of LY2216684 With Alcohol in Healthy Subjects
Brief Title: A Study of LY2216684 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12613; H9P-EW-LNCV (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Alcoholic Beverages

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY, Alc, Pl-Match Alc, Then Pl-Match LY, Alc, Pl-Match Alc (Experimental): Period 1: 18 milligrams (mg) LY2216684 (LY) administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of an alcoholic (Alc) beverage (with an alcohol dose of 0.6 grams per kilograms [g/kg] for women and 0.7 g/kg for men), taken orally, one time. On Day 8, participants were administered 2 cups of a placebo-matching (Pl-Match) alcoholic beverage, taken orally, one time.
  Period 2: Placebo-matching LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men), taken orally, one time. On Day 8, participants were administered 2 cups of a placebo-matching alcoholic beverage, taken orally, one time.
  There was a 7-day washout period between Periods 1 and 2.
  Interventions: Drug: LY2216684; Drug: Placebo-matching LY2216684; Drug: Placebo-matching alcoholic beverage; Drug: Alcoholic beverage
- Pl-Match LY, Alc, Pl-Match Alc, Then LY, Alc, Pl-Match Alc (Experimental): Period 1: Placebo-matching LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men), taken orally, one time. On Day 8, participants were administered 2 cups of a placebo-matching alcoholic beverage, taken orally, one time.
  Period 2: 18 mg LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men), taken orally, one time. On Day 8, participants were administered 2 cups of a placebo-matching alcoholic beverage, taken orally, one time.
  There was a 7-day washout period between Periods 1 and 2.
  Interventions: Drug: LY2216684; Drug: Placebo-matching LY2216684; Drug: Placebo-matching alcoholic beverage; Drug: Alcoholic beverage
- LY, Pl-Match Alc, Alc, Then Pl-Match LY, Pl-Match Alc, Alc (Experimental): Period 1: 18 mg LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of a placebo-matching alcoholic beverage, taken orally, one time. On Day 8, participants were administered 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men), taken orally, one time.
  Period 2: Placebo-matching LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of a placebo-matching alcoholic beverage, taken orally, one time. On Day 8, participants were administered 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men), taken orally, one time.
  There was a 7-day washout period between Periods 1 and 2.
  Interventions: Drug: LY2216684; Drug: Placebo-matching LY2216684; Drug: Placebo-matching alcoholic beverage; Drug: Alcoholic beverage
- Pl-Match LY, Pl-Match Alc, Alc, Then LY, Pl-Match Alc, Alc (Experimental): Period 1: Placebo-matching LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of a placebo-matching alcoholic beverage, taken orally, one time. On Day 8, participants were administered 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men), taken orally, one time.
  Period 2: 18 mg LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of a placebo-matching alcoholic beverage, taken orally, one time. On Day 8, participants were administered 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men), taken orally, one time.
  There was a 7-day washout period between Periods 1 and 2.
  Interventions: Drug: LY2216684; Drug: Placebo-matching LY2216684; Drug: Placebo-matching alcoholic beverage; Drug: Alcoholic beverage

INTERVENTIONS:
Drug: LY2216684 — Administered orally
  Other Names: Edivoxetine
Drug: Placebo-matching LY2216684 — Administered orally
Drug: Placebo-matching alcoholic beverage — Administered orally
Drug: Alcoholic beverage — Administered orally

SUMMARY:
This study will evaluate the pharmacodynamic and pharmacokinetic interaction of LY2216684 with alcohol in healthy participants. This study will run approximately for 34 days.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or female participants, as determined by medical history and physical examination
* Male participants: Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug
* Female participants: Women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug (hormonal methods of contraception, including oral and implantable contraceptives, are not allowed in this study) or women who are not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or due to menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone [FSH] >40 milli-international units/milliliter [mIU/mL])
* Male and female participants: Examples of reliable methods of birth control include double-barrier methods (for example, condom and spermicide) alone or in combination with vasectomy, vasectomized partners, and abstinence.
* Have a body weight >50 kilogram (kg)
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site
* Have normal blood pressure and pulse rate (in sitting position) as determined by the investigator

Exclusion Criteria:

* Are currently enrolled in or have completed or discontinued within the last 30 days from a clinical trial involving an investigational product other than the study drug used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2216684, related compounds or any components of the formulation
* Are persons who have previously received the investigational product in this study or have completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to Screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders that are capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history or show evidence of significant active neuropsychiatric disease or have a history of suicide attempt or ideation
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Participants with a past history of alcohol dependence/abuse
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Women with a positive pregnancy test or women who are lactating
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing or during the study unless deemed acceptable by the investigator and Sponsor's medical monitor, except for influenza vaccinations
* Have donated blood of more than 500 milliliter (mL) within the last month
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption 48 hours prior to each study period and while resident at the Clinical Research Unit (CRU) (except as required per this protocol); (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or are unwilling to adhere to study caffeine restrictions
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment or are unwilling to abstain during the study
* Have a documented or suspected history of glaucoma
* Participants with known or suspected alcohol dehydrogenase deficiency
* Participants who do not drink alcohol and/or are not willing to drink 4 units of alcohol over a 15-minute period
* Participants determined to be unsuitable by the investigator for any reason

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | LY, Alc, Pl-Match Alc, Then Pl-Match LY, Alc, Pl-Match Alc | Pl-Match LY, Alc, Pl-Match Alc, Then LY, Alc, Pl-Match Alc | LY, Pl-Match Alc, Alc, Then Pl-Match LY, Pl-Match Alc, Alc | Pl-Match LY, Pl-Match Alc, Alc, Then LY, Pl-Match Alc, Alc
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | LY, Alc, Pl-Match Alc, Then Pl-Match LY, Alc, Pl-Match Alc | Pl-Match LY, Alc, Pl-Match Alc, Then LY, Alc, Pl-Match Alc | LY, Pl-Match Alc, Alc, Then Pl-Match LY, Pl-Match Alc, Alc | Pl-Match LY, Pl-Match Alc, Alc, Then LY, Pl-Match Alc, Alc
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 6 | 6
Not Completed | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | LY, Alc, Pl-Match Alc, Then Pl-Match LY, Alc, Pl-Match Alc | Pl-Match LY, Alc, Pl-Match Alc, Then LY, Alc, Pl-Match Alc | LY, Pl-Match Alc, Alc, Then Pl-Match LY, Pl-Match Alc, Alc | Pl-Match LY, Pl-Match Alc, Alc, Then LY, Pl-Match Alc, Alc
Started | 7 | 7 | 6 | 6
Completed | 7 | 7 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Overall: Participants received 18 mg LY2216684 or Placebo-matching LY2216684 administered orally, once daily for 8 days during Periods 1 and 2. On Day 6 and on Day 8 of each period, participants were administered either 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men) or placebo-matching alcoholic beverage, taken orally, one time.
  There was a 7-day washout period between Periods 1 and 2.
Arm/Group | Overall
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19
  Black or African American | 8
  Multiple | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 10 Hours in Power of Attention Composite Score
Description: Power of attention is a measure of focused attention and information processing speed; based on the summed reaction times from the simple reaction time, choice reaction time, and digit vigilance tasks. Scores are measured by response latencies, and smaller scores indicate better function. Least squares (LS) means were calculated using mixed model analysis of covariance (ANCOVA) adjusting for predose, sequence, period, day, time, treatment, and treatment*time as fixed effects and participant within sequence and treatment as random effect.
Time Frame: Baseline, 10 hours
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, placebo-matching LY2216684, or placebo-matching alcoholic beverage with evaluable power of attention data.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Groups:
- LY2216684 + Alcohol: 18 mg LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men), taken orally, one time.
- Placebo-matching LY2216684 + Alcohol: Placebo-matching LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of an alcoholic beverage (with an alcohol dose of 0.6 g/kg for women and 0.7 g/kg for men), taken orally, one time.
- LY2216684 + Placebo-matching Alcohol: 18 mg LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of a placebo-matching alcoholic beverage, taken orally, one time.
- Placebo-matching LY2216684 + Placebo-matching Alcohol: Placebo-matching LY2216684 administered orally, once daily for 8 days. On Day 6, participants were administered 2 cups of a placebo-matching alcoholic beverage, taken orally, one time.
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol | Placebo-matching LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 27 | 27 | 27 | 27
minutes | 67.82 [22.01 to 113.63] | 52.77 [7.05 to 98.5] | 20.6 [-25.13 to 66.33] | 6.78 [-39.13 to 52.69]

2. Primary Outcome: Change From Baseline to 10 Hours in Continuity of Attention Composite Score
Description: Continuity of attention is a measure of sustained attention, combining (summed) accuracy and error measures from the choice reaction time and digit vigilance tasks. The number of correct responses (out of 50) for choice reaction time was added to the total number of targets correctly identified (out of 45) digit vigilance minus the number of false alarms (total score of -45 to 95). A high score reflects someone able to keep his/her mind on a single task for a prolonged period. A negative change from baseline reflects impairment compared to baseline.
  LS means were calculated using mixed model ANCOVA adjusting for predose, sequence, period, day, time, treatment, and treatment*time as fixed effects and participant within sequence and treatment as random effect.
Time Frame: Baseline, 10 hours
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, placebo-matching LY2216684, or placebo-matching alcoholic beverage with evaluable continuity of attention data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol | Placebo-matching LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 27 | 27 | 27 | 27
units on a scale | -4.21 [-6.98 to -1.43] | -1.16 [-3.93 to 1.61] | -3.31 [-6.08 to -0.54] | -1.24 [-4 to 1.53]

3. Primary Outcome: Change From Baseline to 10 Hours in Postural Stability
Description: The ability to stand upright without moving was assessed using equipment modeled on the Wright Ataxia-meter. To measure movements, a cord was attached to the participant who was required to stand for one minute, as still as possible, with feet apart and eyes closed. The amount of sway is expressed as the total angular movement calibrated in units of one-third degree of angle of sway.
  The amount of sway is expressed as the total angular movement in the antero-posterior plane and calibrated in units of one-third degree of angle of sway. Higher result indicates better postural stability. A negative change from baseline reflects impairment compared to baseline. LS means were calculated using mixed model ANCOVA adjusting for predose, sequence, period, day, time, treatment, and treatment*time as fixed effects and participant within sequence and treatment as random effect.
Time Frame: Baseline, 10 hours
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, placebo-matching LY2216684, or placebo-matching alcoholic beverage with evaluable postural stability data.
Measure: Least Squares Mean (95% Confidence Interval); unit: 1/3 degree of angle of sway
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol | Placebo-matching LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 27 | 27 | 27 | 27
1/3 degree of angle of sway | 0.14 [-5.38 to 5.66] | -3.51 [-9.03 to 2] | -3.65 [-9.17 to 1.87] | 5.2 [-0.32 to 10.72]

4. Primary Outcome: Change From Baseline to 10 Hours in Self-Rated Alertness
Description: Assessed via the Bond and Lader Visual Analogue Scale (VAS), which utilizes a 16-point scale of 0 to 100 with 0 representing the worst rating and 100 representing the best rating. LS means were calculated using mixed model ANCOVA adjusting for predose, sequence, period, day, time, treatment, and treatment*time as fixed effects and participant within sequence and treatment as random effect.
Time Frame: Baseline, 10 hours
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, placebo-matching LY2216684, or placebo-matching alcoholic beverage with evaluable self-rated alertness data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol | Placebo-matching LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 27 | 27 | 27 | 27
units on a scale | 3.85 [-4.25 to 11.95] | -2.37 [-10.47 to 5.72] | 11.88 [3.77 to 19.98] | 3.02 [-5.1 to 11.14]

5. Secondary Outcome: Pharmacokinetics: Observed Maximum Plasma Concentration (Cmax) of LY2216684
Time Frame: Predose through 24 hours postdose
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, or placebo-matching alcoholic beverage with evaluable LY2216684-concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliters (ng/mL)
Arm/Group | LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 27 | 27
nanograms/milliliters (ng/mL) | 60.2 (39) | 58.0 (36)

6. Secondary Outcome: Pharmacokinetics: Observed Cmax of Alcohol
Time Frame: Predose through 24 hours postdose
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, or placebo-matching LY2216684 with evaluable alcohol-concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimoles/liters (mmol/L)
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol
Number analyzed (Participants) | 27 | 27
millimoles/liters (mmol/L) | 11.4 (30) | 13.8 (22)

7. Secondary Outcome: Pharmacokinetics: Observed Time to Maximum Plasma Concentration (Tmax) of LY2216684
Time Frame: Predose through 24 hours postdose
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 26 | 26
hours | 4.00 [1.85 to 5.92] | 2.94 [1.08 to 5.92]

8. Secondary Outcome: Pharmacokinetics: Observed Tmax of Alcohol
Time Frame: Predose through 24 hours postdose
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol
Number analyzed (Participants) | 26 | 26
hours | 0.92 [0.50 to 1.92] | 0.92 [0.50 to 1.92]

9. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve Over a Dosing Interval (AUCt) of LY2216684
Time Frame: Predose through 24 hours postdose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliters (ng*h/mL)
Arm/Group | LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 26 | 27
nanograms*hours/milliliters (ng*h/mL) | 717 (41) | 678 (38)

10. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve From Time Zero to the Last Time Point With a Measurable Concentration (AUC[0-tlast]) of Alcohol
Time Frame: Predose through 12 hours postdose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimoles*hours/liters (mmol*h/L)
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol
Number analyzed (Participants) | 27 | 27
millimoles*hours/liters (mmol*h/L) | 29.7 (49) | 34.5 (43)

11. Secondary Outcome: Change From Baseline to 1, 2, 3, 4.5, 6, 8, and 10 Hours in Working Memory
Description: Working memory is a sum of accuracy measures from the numeric and spatial working memory tasks known as the sensitivity index (SI). Working Memory SI is based on how fast the participant responds correctly and how many are correct responses. SI ranging from zero (chance performance) to one (perfect accuracy). A high score reflects someone able to hold in memory for a prolonged period. A negative change from baseline reflects impairment compared to baseline.
  A series of 5 digits were presented on a computer screen, every second, for the participant to hold in memory. Followed by 30 probe digits, the participant had to decide whether it appeared in the original series by responding with 'Yes' or 'No'. This was repeated 2 times using different series and probes.
  LS mean was calculated using mixed model ANCOVA adjusting for predose, sequence, period, day, time, treatment, and treatment*time as fixed effects and participant within sequence and treatment as random effect.
Time Frame: Baseline, 1, 2, 3, 4.5, 6, 8, and 10 hours
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, placebo-matching LY2216684, or placebo-matching alcoholic beverage with evaluable working memory data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol | Placebo-matching LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 27 | 27 | 27 | 27
Units on a scale
  Hour 1 | -0.12 [-0.2 to -0.03] | -0.12 [-0.21 to -0.04] | -0.1 [-0.19 to -0.02] | -0.02 [-0.1 to 0.07]
  Hour 2 | -0.27 [-0.42 to -0.12] | -0.29 [-0.44 to -0.14] | -0.13 [-0.28 to 0.02] | -0.12 [-0.27 to 0.03]
  Hour 3 | -0.2 [-0.34 to -0.07] | -0.18 [-0.31 to -0.05] | -0.06 [-0.19 to 0.08] | -0.04 [-0.17 to 0.09]
  Hour 4.5 | -0.15 [-0.29 to -0.01] | -0.11 [-0.25 to 0.03] | -0.2 [-0.34 to -0.06] | -0.2 [-0.35 to -0.06]
  Hour 6 | -0.1 [-0.2 to -0.01] | -0.09 [-0.19 to 0.01] | -0.06 [-0.16 to 0.03] | -0.07 [-0.17 to 0.02]
  Hour 8 | -0.03 [-0.15 to 0.08] | -0.05 [-0.17 to 0.06] | -0.08 [-0.19 to 0.04] | -0.13 [-0.24 to -0.01]
  Hour 10 | -0.21 [-0.35 to -0.07] | -0.09 [-0.23 to 0.06] | -0.16 [-0.3 to -0.01] | -0.06 [-0.21 to 0.08]

12. Secondary Outcome: Change From Baseline to 1, 2, 3, 4.5, 6, 8, and 10 Hours in Episodic Memory
Description: Episodic memory is based on how accurate the participant responds using the measures from immediate word recall (range 0-15), delayed word recall (range 0-15), word recognition (range 0-15), and picture recognition (range 0-20) tasks. The sum of four the accuracy scores, are summed, and averaged to provide a composite score (range 0-37.5). This composite score reflects the ability to store, hold, and retrieve information of an episodic nature (such as an event, a name, an object, a scene, or an appointment). A high score reflects someone able to recall memory for a prolonged period. A negative change from baseline reflects impairment compared to baseline.
  LS mean was calculated using mixed model ANCOVA adjusting for predose, sequence, period, day, time, treatment, and treatment*time as fixed effects and participant within sequence and treatment as random effect.
Time Frame: Baseline, 1, 2, 3, 4.5, 6, 8, and 10 hours
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, placebo-matching LY2216684, or placebo-matching alcoholic beverage with evaluable episodic memory data.
Measure: Geometric Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol | Placebo-matching LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 27 | 27 | 27 | 27
units on a scale
  Hour 1: number analyzed (Participants) | 27 | 27 | 26 | 27
  Hour 1 | -29.13 [-45.64 to -12.62] | -30.56 [-47.05 to -14.07] | -24.81 [-41.57 to -8.05] | -19.29 [-35.81 to -2.77]
  Hour 2 | -96.35 [-115.59 to -77.11] | -97.54 [-116.76 to -78.32] | -44.3 [-63.53 to -25.07] | -41.64 [-60.88 to -22.39]
  Hour 3 | -76.72 [-93.96 to -59.48] | -74.27 [-91.49 to -57.04] | -34.92 [-52.15 to -17.69] | -30.58 [-47.84 to -13.33]
  Hour 4.5 | -65.06 [-82.57 to -47.55] | -52.23 [-69.73 to -34.74] | -50.78 [-68.28 to -33.28] | -34.29 [-51.81 to -16.77]
  Hour 6 | -39.56 [-56.48 to -22.65] | -49.7 [-66.6 to -32.8] | -41.34 [-58.24 to -24.43] | -38.86 [-55.78 to -21.93]
  Hour 8 | -42.28 [-58.63 to -25.93] | -43.65 [-59.98 to -27.32] | -46.09 [-62.43 to -29.75] | -35.95 [-52.31 to -19.6]
  Hour 10 | -46.78 [-65.31 to -28.26] | -34.33 [-52.84 to -15.82] | -41.95 [-60.47 to -23.44] | -39.04 [-57.58 to -20.5]

13. Secondary Outcome: Change From Baseline to 1, 2, 3, 4.5, 6, 8, and 10 Hours in Speed of Retrieval of Information From Memory
Description: Speed of retrieval is a measure of complex information processing speed, summing reaction times from the two working memory (numeric and spatial) tasks and the two episodic recognition (word recognition and picture recognition) tasks. This composite score reflects the time it takes to decide correctly whether an item is held in working memory or episodic secondary memory.Scores are measured by response latencies, and smaller scores indicate better function. A negative change from baseline reflects impairment compared to baseline.
  LS means calculated using mixed model ANCOVA adjusting for predose, sequence, period, day, time, treatment, and treatment*time as fixed effects and participant within sequence and treatment as random effect.
Time Frame: Baseline, 1, 2, 3, 4.5, 6, 8, and 10 hours
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, placebo-matching LY2216684, or placebo-matching alcoholic beverage with evaluable speed of retrieval of information from memory data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millisecond (msec)
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol | Placebo-matching LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 27 | 27 | 27 | 27
millisecond (msec)
  Hour 1: number analyzed (Participants) | 27 | 27 | 26 | 27
  Hour 1 | -38.46 [-198.46 to 121.55] | 36.22 [-123.97 to 196.4] | 42.51 [-118.79 to 203.8] | 138.87 [-21.27 to 299.02]
  Hour 2 | 104.48 [-199.46 to 408.42] | 316.09 [12.06 to 620.12] | 59.65 [-244.29 to 363.59] | 197.37 [-106.64 to 501.38]
  Hour 3 | 43.69 [-215.33 to 302.7] | 283.63 [24.51 to 542.75] | 51.53 [-207.49 to 310.54] | 24.55 [-234.55 to 283.65]
  Hour 4.5 | 30.12 [-219.38 to 279.62] | 61.93 [-187.69 to 311.54] | -121.55 [-371.06 to 127.96] | 169.34 [-80.26 to 418.93]
  Hour 6 | -116.69 [-266.39 to 33.01] | 46.44 [-103.45 to 196.33] | -90.46 [-240.16 to 59.25] | -114.87 [-264.72 to 34.98]
  Hour 8 | -116.72 [-315.54 to 82.11] | -48.13 [-247.09 to 150.84] | 55.62 [-143.21 to 254.45] | -120.29 [-319.23 to 78.64]
  Hour 10 | -74.78 [-233.06 to 83.49] | -136.62 [-295.08 to 21.83] | -108.12 [-266.4 to 50.17] | -129.8 [-288.22 to 28.61]

14. Secondary Outcome: Change From Baseline to 1, 2, 3, 4.5, 6, 8, and 10 Hours in Self-Ratings of Calmness and Contentment
Description: as for outcome 4
Time Frame: Baseline, 1, 2, 3, 4.5, 6, 8, and 10 hours
Population: Participants who received at least one dose of LY2216684, alcoholic beverage, placebo-matching LY2216684, or placebo-matching alcoholic beverage with evaluable calmness and contentment self-ratings.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol | LY2216684 + Placebo-matching Alcohol | Placebo-matching LY2216684 + Placebo-matching Alcohol
Number analyzed (Participants) | 27 | 27 | 27 | 27
units on a scale
  Self-rated Alertness, Hour 1: number analyzed (Participants) | 27 | 27 | 26 | 27
  Self-rated Alertness, Hour 1 | 2.98 [-4.18 to 10.14] | 4.57 [-2.59 to 11.73] | 3.64 [-3.63 to 10.91] | 6.06 [-1.13 to 13.25]
  Self-rated Alertness, Hour 2 | 17.09 [8.81 to 25.37] | 14.08 [5.8 to 22.36] | 0.76 [-7.53 to 9.06] | 3.64 [-4.67 to 11.94]
  Self-rated Alertness, Hour 3 | 23.67 [15.05 to 32.3] | 26.25 [17.63 to 34.87] | 9.04 [0.41 to 17.67] | 1.22 [-7.42 to 9.87]
  Self-rated Alertness, Hour 4.5 | 27.19 [17.76 to 36.61] | 20.74 [11.32 to 30.16] | 16.26 [6.83 to 25.69] | 9.82 [0.37 to 19.26]
  Self-rated Alertness, Hour 6 | 23.66 [13.93 to 33.39] | 17.25 [7.52 to 26.98] | 15.13 [5.4 to 24.87] | 7.55 [-2.2 to 17.3]
  Self-rated Alertness, Hour 8 | 12.69 [3.75 to 21.63] | 3.63 [-5.31 to 12.57] | 12.38 [3.43 to 21.33] | 3.03 [-5.93 to 11.99]
  Self-rated Alertness, Hour 10 | 3.85 [-4.25 to 11.95] | -2.37 [-10.47 to 5.72] | 11.88 [3.77 to 19.98] | 3.02 [-5.1 to 11.14]
  Self-rated Contentment, Hour 1: number analyzed (Participants) | 27 | 27 | 26 | 27
  Self-rated Contentment, Hour 1 | 3.28 [-0.98 to 7.55] | 0.95 [-3.32 to 5.22] | 2.77 [-1.57 to 7.11] | 4.34 [0.07 to 8.6]
  Self-rated Contentment, Hour 2 | 3.72 [-2.72 to 10.16] | 1.5 [-4.95 to 7.95] | 1.64 [-4.81 to 8.09] | 2.79 [-3.65 to 9.23]
  Self-rated Contentment, Hour 3 | 8.41 [2.05 to 14.77] | 7.12 [0.75 to 13.49] | 5.69 [-0.67 to 12.06] | 1.32 [-5.05 to 7.68]
  Self-rated Contentment, Hour 4.5 | 16.98 [8.97 to 24.99] | 8.5 [0.49 to 16.51] | 11.39 [3.38 to 19.4] | 5.03 [-2.98 to 13.03]
  Self-rated Contentment, Hour 6 | 18.14 [9.12 to 27.17] | 10.85 [1.82 to 19.88] | 10.68 [1.65 to 19.71] | 4.57 [-4.45 to 13.6]
  Self-rated Contentment, Hour 8 | 9.97 [2.14 to 17.79] | 0.98 [-6.85 to 8.81] | 9.68 [1.86 to 17.51] | 2.7 [-5.12 to 10.53]
  Self-rated Contentment, Hour 10 | 2.47 [-5.14 to 10.07] | 0.44 [-7.17 to 8.05] | 10.16 [2.55 to 17.77] | 3.72 [-3.89 to 11.32]

ADVERSE EVENTS:
Groups:
- LY2216684 + Placebo-matching Alcohol: 18 mg LY2216684 administered orally, once daily for 8 days. On Day 8, participants were administered 2 cups of a placebo-matching (Pl-Match) alcoholic beverage, taken orally, one time.
- Placebo-matching LY2216684 + Placebo-matching Alcohol: Placebo-matching LY2216684 administered orally, once daily for 8 days. On Day 8, participants were administered 2 cups of a placebo-matching (Pl-Match) alcoholic beverage, taken orally, one time.
Arm/Group | LY2216684 + Placebo-matching Alcohol | Placebo-matching LY2216684 + Placebo-matching Alcohol | LY2216684 + Alcohol | Placebo-matching LY2216684 + Alcohol
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 16/27 | 8/27 | 10/27 | 8/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 + Placebo-matching Alcohol (N=27) | Placebo-matching LY2216684 + Placebo-matching Alcohol (N=27) | LY2216684 + Alcohol (N=27) | Placebo-matching LY2216684 + Alcohol (N=27)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (5) | 3 (3) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 4 (5) | 1 (2) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/10 (1) | 0/10 (0) | 0/10 (0) | 0/10 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/10 (0) | 0/10 (0) | 1/10 (1) | 0/10 (0)
Pelvic pain (Reproductive system and breast disorders) | 0/10 (0) | 0/10 (0) | 1/10 (1) | 0/10 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days